CLINICAL TRIAL: NCT07058350
Title: Association Between Radiological Stenosis Level and Patient Questionnaires in Patients With Lumbar Spinal Stenosis: A Cross-Sectional Study
Brief Title: Radiological Lumbar Spinal Stenosis Level and Patient Questionnaires
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Selda Çiftci, Medical Doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 04.08.2025/approval no:4828
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-06

CONDITIONS: Lumbar Spinal Stenosis; Low Back Pain
Keywords: lumbar spinal stenosis; low back pain; İstanbul low back pain disability index; Oswestry Disability Index; Swiss Spinal Stenosis Questionnaire
MeSH Terms: conditions — Spinal Stenosis; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Those with radiological lumbar spinal stenosis: Those with Grade 1 or 2 or 3 according to the Lee radiological spinal stenosis staging system
- Those without radiological lumbar spinal stenosis: Those with Grade 0 according to the Lee radiological spinal stenosis staging system

SUMMARY:
One of the important causes of low back pain is lumbar spinal stenosis. With the increasing prevalence of magnetic resonance imaging (MRI), lumbar spinal stenosis grading systems have been developed. The Lee and Schizas lumbar spinal stenosis grading systems are widely used. Patient questionnaires are also used especially in treatment follow-ups. This study aimed to compare the compliance of patient questionnaires with the presence or absence of radiological stenosis and the degree of stenosis if present.

DETAILED DESCRIPTION:
Patients who apply to our Physical Medicine and Rehabilitation out-patient clinic with complaints of low back pain and who have or do not have lumbar spinal stenosis on lumbar spinal MRI will be screened. Demographic values, accompanying diseases, radiological staging of lumbar spinal stenosis, Oswestry Disability Index, Istanbul Low Back Pain Disability Questionnaire, Swiss Spinal Stenosis Questionnaire will be evaluated. Pain levels will be evaluated with Visual Analog Scale (VAS). Radiological stenosis level will be determined with Lee radiological spinal stenosis classification system. Those with and without stenosis will be determined. In addition, subgroup analysis will be performed by creating subgroups with mild, moderate and severe stenosis in the stenosis group. Evaluations will be made at the L4-L5 vertebrae level, where degenerative spinal stenosis is most frequently seen. All questionnaires will be filled in both groups with and without stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 and over with low back pain
* Those who have had a lumbar magnetic resonance imaging (MRI) scan within the last year

Exclusion Criteria:

* Patients with congenital lumbar spinal stenosis
* Patients with traumatic lumbar spinal stenosis
* Patients with iatrogenic lumbar spinal stenosis
* Those with a history of lumbar vertebral surgery
* Those with cognitive impairment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 50 and over with low back pain
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | Day 1
  The Oswestry Disability Index (ODI) is used to measure the degree of functional limitations caused by pain in patients with low back pain. The questionnaire provides the user with detailed information about the general daily functioning of a patient with low back pain. Questions are included regarding pain intensity, self-care, lifting, moving, sitting or standing, sleeping, sexual life, social life, and travel/transportation. A score of 0 indicates no limitations due to pain, while a score of 5 indicates the greatest perceived limitation in an activity due to pain. It is calculated by dividing the total score by the score range and multiplying the result by 100 to obtain the percentage value of the index. 0% indicating no disability and 100% indicating the highest level of disability.
İstanbul Low Back Pain Disability Questionnaire | Day 1
  The Istanbul Low Back Pain Disability Index consists of 18 questions that evaluate the effects of low back pain on activities such as going up and down stairs, walking, bathing, brushing teeth, dressing, etc. If a person can do it "without any difficulty", 0 points, if "with little difficulty", 1 point, if "with some difficulty", 2 points, if "with great difficulty", 3 points, if "almost impossible", 4 points, and "impossible" (5 points) are used to obtain a total score of 0-90. A total score of 0 indicates no disability, while 90 indicates maximum disability.
Swiss Spinal Stenosis Questionnaire | Day 1
  The Swiss Spinal Stenosis Questionnaire consists of 18 questions. The first 7 questions concern the patient's symptoms. The first three questions concern pain (intensity, frequency and back pain) and the last four questions concern neuroischemic symptoms (numbness or tingling, weakness and balance disorders). Each question is scored from 1 to 5 (maximum 35 points). The next 5 questions concern the patients' physical activity and each question is scored from 1 to 4 (maximum 20 points). A higher score indicates a more severe disease. The last 6 questions concern the patients' satisfaction with surgical treatment and each is scored from 1 to 4. A higher score indicates less satisfaction with surgery.

SECONDARY OUTCOMES:
Visual Analog Scale | Day 1
  Using a ruler, the score is determined by measuring the distance (mm) on the 10 cm line between the "no pain" anchor and the patient's mark, providing a score range of 0-100. A higher score indicates greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Kuran, Professor, Medical Doctor, Study Director — Şişli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided